CLINICAL TRIAL: NCT05345171
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Adeno-associated Virus (AAV) Serotype 8 (AAV8)-Mediated Gene Transfer of Human Ornithine Transcarbamylase (OTC) in Patients With Late-onset OTC Deficiency
Brief Title: Clinical Study of DTX301 AAV-Mediated Gene Transfer for Ornithine Transcarbamylase (OTC) Deficiency
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTX301-CL301; 2020-003384-25 (EudraCT Number); 2024-514337-38-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: OTC Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease | interventions — Adrenal Cortex Hormones; Prednisolone; Sodium Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DTX301 (Experimental): Participants receive single peripheral intravenous (IV) infusion of DTX301 in solution. Between Week 36 and Week 64, participants may receive single peripheral IV infusion of placebo.
  Interventions: Genetic: DTX301; Other: Placebo; Drug: Oral Corticosteroids; Drug: Placebo for oral corticosteroids; Drug: Sodium Acetate
- Placebo, Then DTX301 (Experimental): Participants receive single peripheral IV infusion of placebo. Between Week 36 and Week 64, participants receive single peripheral IV infusion of DTX301 in solution.
  Interventions: Genetic: DTX301; Other: Placebo; Drug: Oral Corticosteroids; Drug: Placebo for oral corticosteroids; Drug: Sodium Acetate

INTERVENTIONS:
Genetic: DTX301 — non-replicating, self-complementary recombinant adeno-associated virus serotype 8 (AAV8) vector
  Other Names: avalotcagene ontaparvovec
Other: Placebo — normal saline infusion
Drug: Oral Corticosteroids — Participants who receive DTX301 solution will receive oral corticosteroids.
  Other Names: Prednisolone
Drug: Placebo for oral corticosteroids — Participants who receive Placebo will receive placebo corticosteroids to maintain the study blind
Drug: Sodium Acetate — A tracer for the Ureagenesis Rate Test (URT)

SUMMARY:
The primary objective is to evaluate the efficacy of DTX301 on the improvement of ornithine transcarbamylase (OTC) function by maintaining safe plasma ammonia levels.

DETAILED DESCRIPTION:
This study is a Phase 3, randomized, double-blind, placebo-controlled study of DTX301 in patients with late-onset OTC deficiency 12 years of age and older.

Participants will be randomized 1:1 to DTX301 or placebo and followed closely for 36-64 weeks. Between Week 36 and Week 64, eligible participants will cross over and receive DTX301 if they had previously received placebo, and some who received DTX301 may receive placebo.

The planned study duration is up to 324 weeks. Upon completion of this study or early withdrawal, all participants who received DTX301 are invited to enroll in the Disease Monitoring Program (DMP) for follow-up for up to an additional 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed clinical diagnosis of late-onset OTC deficiency with historical documentation by enzymatic (ie, liver biopsy), biochemical (ie, hyperammonemia in the presence of elevated plasma glutamine, low citrulline, and elevated spot urine orotic acid), or molecular testing (ie, OTC analysis)
* Free from symptomatic hyperammonemia and has not required emergent active intervention for hyperammonemia within 4 weeks before screening/baseline
* If on ongoing daily ammonia scavenger therapy, must be at stable daily dose(s) for ≥ 4 weeks prior to screening
* If on a protein-restricted diet, must be on a stable total daily protein intake that does not vary more than 20% for ≥ 4 weeks prior to screening
* From the time written informed consent through Visit 28, females of childbearing potential and fertile males must consent to use highly effective contraception. If female, agree not to become pregnant. If male, agree not father a child or donate sperm

Key Exclusion Criteria:

* Significant hepatic inflammation or cirrhosis
* Estimated glomerular filtration rate < 60 mL/min/1.73 m2 at screening by the 2021 CKD-EPI creatinine-based formula (Inker et al., 2021) for patients ≥ 18 years of age or the Schwartz bedside formula (Schwartz and Work, 2009) for patients < 18 years of age
* Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, documented by current use of antiviral therapy for HBV or HCV or by hepatitis B surface antigen (HBsAg) or HCV RNA positivity
* Active infection (viral or bacterial)
* Detectable pre-existing antibodies to the AAV8 capsid
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results
* Participation (current or previous) in another gene transfer study

Note: Additional inclusion/exclusion criteria may apply, per protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Plasma Ammonia as Measured by 24-Hour Ammonia (AUC0-24) | Week 36
Complete Responder Rate at the Final Study Visit After DTX301 Exposure | Up to 64 Weeks Post DTX301 Infusion

SECONDARY OUTCOMES:
Percentage of Complete Responders or Responders After DTX301 Exposure | Up to 64 Weeks Post DTX301 Infusion
Annualized Event Rate of Hyperammonemic Crises (HACs) Pre-DTX301 Exposure vs Post-DTX301 Exposure | Pre-enrollment, Baseline, Up to 64 Weeks Post DTX301 Infusion
Annualized Event Rate of Interim Clinical Events (ICEs) Pre-DTX301 Exposure vs Post-DTX301 Exposure | Pre-enrollment, Baseline, Up to 64 Weeks Post DTX301 Infusion
Change from Baseline in Plasma Ammonia (AUC0-24) | Baseline, Up to Week 36
Change in Plasma Ammonia (AUC0-24) After DTX301 Exposure | Up to 64 Weeks Post DTX301 Infusion
Percentage of Participants Who Have Achieved Complete Management Response (CMR) or Management Response (MR) After DTX301 Exposure | Up to 64 Weeks Post DTX301 Infusion
Change in Baseline Disease Management (Dietary Protein and Total Scavenger Medication Use) With Plasma Ammonia (AUC0-24) | Up to 64 Weeks Post DTX301 Infusion
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs, Related Serious TEAEs and Adverse Events of Special Interest (AESIs) | Up to Week 324
Number of Participants With Anti-OTC Antibodies | Up to Week 324
Long-Term Durability of Response | Up to 64 Weeks Post DTX301 Infusion
  Based Upon Number of Complete Responders or Responders That Have ≥ 2 Consecutive Visits as a Complete Responder or Responder and Do Not Return to a Lower Responder Status for > 1 Consecutive Visit
Change in Plasma Ammonia (AUC0-24) for Participants Who Have an Elevated Ammonia AUC0-24 at Baseline | Baseline, Up to 64 Weeks Post DTX301 Infusion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (16):
- United States (4):
  - University of California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- The Hospital for Sick Children, Toronto, Ontario, Canada
- France (2):
  - Hopital Femme Mere Enfant, Bron
  - Necker-Enfants Maladas Hospital, Paris
- Universitatsklinikum Heidelberg, Heidelberg, Germany
- Japan (2):
  - Kumamoto University Hospital, Kumamoto
  - Fujita Health University Hospital, Toyoake
- Erasmus Universitair Medisch Centrum Rotterrdam, Rotterdam, Netherlands
- Centro Hospitalar Universitario de Sao Joao, Porto, Portugal
- Fundacio Hospital Universitari Vall D'Hebron-Institute de Recerca, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baruteau J, Brunetti-Pierri N, Gissen P. Liver-directed gene therapy for inherited metabolic diseases. J Inherit Metab Dis. 2024 Jan;47(1):9-21. doi: 10.1002/jimd.12709. Epub 2024 Jan 3. PMID 38171926
- See also: Ultragenyx Patient Advocacy/OTC Disease Information — https://ultrarareadvocacy.com/conditions-we-study/ornithine-transcarbamylase-otc-deficiency/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/